CLINICAL TRIAL: NCT02108041
Title: Medical Decision-Making in a Virtual Clinical Setting
Brief Title: Personalized Medicine Decision-Making in a Virtual Clinical Setting
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914075; 14-HG-N075
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-10-17

CONDITIONS: Deep Vein Thrombosis; Blood Clots
Keywords: Physicians; Genomics; Internal Medicine; Warfarin; Natural History
MeSH Terms: conditions — Venous Thrombosis; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Physicians that interact with the black/High SES avatar patien: Medical residents will then be randomized to be exposed to a virtual patient with one of 4 race/SES profiles, this one being a female patient who is Upper-Middle Income and Black/African American.
- Physicians that interact with the black/Low SES avatar patient: Medical residents will then be randomized to be exposed to a virtual patient with one of 4 race/SES profiles, this one being a female patient who is low-Middle Income and Black/African American.
- Physicians that interact with the white race/high SES avatar: Medical residents will then be randomized to be exposed to a virtual patient with one of 4 race/SES profiles, this one being a female patient who is Upper-Middle Income White andCaucasian.
- Physicians that interact with the white race/low SES avatar p: Medical residents will then be randomized to be exposed to a virtual patient with one of 4 race/SES profiles, this one being a female patient who is low Income White and Caucasian.

SUMMARY:
Background:

-How people respond to drugs depends in part on their genes. For some drugs, doctors can use an individuals genetic background to help in dosing the drug. Researchers want to know how doctors incorporate personalized or genomic medicine into clinical practice.

Objective:

-To study how physicians make personalized treatment decisions

Eligibility:

-Healthy adult primary care physicians who are internal (or family) medicine residents.

Design:

* Participants will complete a screening form.
* Participants will put on a headset, called a head-mounted display, showing a virtual reality environment.
* The environment will contain an exam room and the virtual patient.
* After interacting with the virtual patient, participants will complete a series of survey measures.
* Participation will last for about 60 minutes. The virtual patient interaction and follow-up questions will be audio taped.

DETAILED DESCRIPTION:
This study will examine factors related to primary care physicians clinical decision-making. Using a virtual clinical interaction experiment, we aim to better understand physicians decision-making processes and to explore their communication behaviors toward patients in the clinical encounter. Physician participants will enter a virtual exam room where they will be asked to respond to a virtual patient, acting as her primary care physician in a follow-up visit to evaluate her for depression. Various aspects of physician communication in the virtual clinic and self-report measures related to decision-making will be analyzed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All physicians will be healthy adult volunteers who are medical residents in the internal medicine specialty.

EXCLUSION CRITERIA:

1. persons with seizure or vestibular disorders;
2. persons who are highly prone to motion sickness;
3. those without normal or normal to corrected vision or hearing;
4. all current and past employees and contractors of NHGRI; and
5. persons who have received information about the study purpose or procedure from a past participant.

NHGRI employees are excluded for this protocol because they are likely to have specialized genomic knowledge and may think differently about genomics in the clinical interaction.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Internal medicine and family medicine residents will be recruited from diverse national sites for the study, and the virtual reality environment will be brought to them through the use of a head-mounted display and laptop
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
To explore how physicians use genetic testing for anticoagulant (warfarin) dosage in patients of different racial/ethnic and SES backgrounds | Outcome measurements are assessed on the same date of the study visit.
  To explore how physicians use genetic testing for anticoagulant (warfarin) dosage in patients of different racial /ethnic and SES backgrounds

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (5):
- United States (5):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Harvard School of Public Health, Boston, Massachusetts
  - Michigan State University, Flint, Michigan
  - Columbia University, New York, New York
  - University of Oregon, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No
We will provide data contingent on special requests form other researchers.

REFERENCES:
- [Background] Green AR, Carney DR, Pallin DJ, Ngo LH, Raymond KL, Iezzoni LI, Banaji MR. Implicit bias among physicians and its prediction of thrombolysis decisions for black and white patients. J Gen Intern Med. 2007 Sep;22(9):1231-8. doi: 10.1007/s11606-007-0258-5. Epub 2007 Jun 27. PMID 17594129
- [Background] Armstrong K. Genomics and health care disparities: the role of statistical discrimination. JAMA. 2012 Nov 21;308(19):1979-80. doi: 10.1001/2012.jama.10820. No abstract available. PMID 23138130